CLINICAL TRIAL: NCT04464434
Title: Upfront Autologous Hematopoietic Stem Cell Transplantation Versus Immunosuppressive Medication in Early Diffuse Cutaneous Systemic Sclerosis: an International Multicentre, Open-label, Randomized Con-trolled Trial
Brief Title: Upfront Autologous HSCT Versus Immunosuppression in Early Diffuse Cutaneous Systemic Sclerosis
Acronym: UPSIDE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Boehringer Ingelheim (Industry); Miltenyi Biotec, Inc. (Industry)
Responsible Party: Principal Investigator, Jacob M van Laar, Principal Investigator, Clinical professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL72607.041.20
Record Dates: First submitted 2020-06-25; First posted 2020-07-09 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Systemic Sclerosis; Systemic Scleroses, Diffuse; Scleroderma; Scleroderma, Diffuse; Autologous Stem Cell Transplantation; Cyclophosphamide; Mycophenolate Mofetil; Treatment Strategy
Keywords: Randomized controlled trial; Autologous stem cell transplantation; Systemic Sclerosis; Cyclophosphamide; Mycophenolate Mofetil; Upfront; Treatment strategy; Event Free survival
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Intervention Model Description: This multicentre, randomized, open label trial aims to compare two treatment strategies in early dcSSc: upfront autologous HSCT versus i.v. CYC pulse therapy followed by MMF and HSCT as rescue option.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upfront autologous HSCT (Experimental)
  Interventions: Procedure: Upfront autologous HSCT
- Immunosuppressive therapy (Active Comparator): 12 monthly i.v. pulses CYC 750 mg/m2 (= 9 g/m2 cumulative) followed by at least 12 months of oral MMF daily (3 grams as maximum daily dosage) or mycophenolic acid (up to 2.160 grams daily).
  Hyperhydration, alkalinisation of the urine and mesna is recommended, and will be given according to local protocols in order to prevent haemorrhagic cystitis.
  Interventions: Procedure: Upfront autologous HSCT

INTERVENTIONS:
Procedure: Upfront autologous HSCT — HSCT comprises the following consecutive steps:
  1. Mobilisation
     * Infusions of CYC 2g/m2 on 1 day.
     * Hyperhydration, alkalinisation of urine and mesna to prevent haemorrhagic cystitis.
     * Filgrastim (G-CSF) 5-10 μg/kg/day subcutaneously for 5 days (or more when necessary).
  2. Leukapheresis Prompt start of leukapheresis is required at a CD34+ cell count of ≥10-20/μL. Goal: at least 2 x 10^6 CD34+ cells per kilogram body weight.
  3. Conditioning
     * CYC 50 mg/kg/day intravenously for 4 consecutive days (total 200 mg/kg)
     * Rabbit Antithymocyte Globulin (rbATG), a total dose of 7.5 mg/kg i.v., from Genzyme.
     Hyperhydration, alkalinisation of the urine and mesna will be given to prevent haemorrhagic cystitis.
     I.v. methylprednisolone 2 mg/kg will be administered on the days ATG, to improve tolerability of the ATG.
  4. Peripheral stem cell infusion The number of CD34+ cells to be reinfused should be ≥ 2.0 x 10^6/kg.

SUMMARY:
HSCT has been implemented in (inter)national treatment guidelines for diffuse cutaneous systemic sclerosis (dcSSc) and is offered in clinical care and reimbursed by national health insurance in several European countries. However, data and specific guidelines on the best timing of HSCT in the course of dcSSc are lacking. In particular, it is unclear whether HSCT should be positioned as upfront therapy or as rescue treatment for patients not responding to conventional immunosuppressive therapy.

This multicentre, randomized, open label trial aims to compare two treatment strategies used in usual care: upfront autologous HSCT versus usual care with (intravenous (i.v.) cyclophosphamide (CYC) pulse therapy followed by mycophenolate mofetil (MMF) and HSCT as rescue option).

DETAILED DESCRIPTION:
Rationale: This multicentre, randomized, open label trial aims to compare two treatment strategies used in usual care: upfront autologous HSCT versus usual care with (intravenous (i.v.) cyclophosphamide (CYC) pulse thera-py followed by mycophenolate mofetil (MMF) and HSCT as rescue option). HSCT has been implemented in (inter)national treatment guidelines for diffuse cutaneous systemic sclerosis (dcSSc) and is offered in clinical care and reimbursed by national health insurance in several European countries. However, data and specific guidelines on the best timing of HSCT in the course of dcSSc are lacking.

In particular, it is unclear whether HSCT should be positioned as upfront therapy or as rescue treatment for patients not responding to conventional im-munosuppressive therapy. Given the risks and costs associated with HSCT, it may be preferable to evaluate the patient's response to immunosuppressive therapy before proceeding to HSCT. Considering HSCT as a rescue treatment could significantly delay the need for a potentially harmful treatment and may be an efficient approach from a health economic perspective as HSCT is a highly specialized, resource intensive and expensive medical procedure. On the other hand, in the time frame needed to evaluate the effect of immunosuppressive therapy, pulmonary and cardiac involvement may develop, negatively influencing a patient's prognosis and possibly leading to a contra-indication for HSCT. We hypothesize that upfront HSCT results in less toxicity and medical costs in the long run. Therefore, we propose a multicentre randomized open label trial in chemotherapy naive patients with early dcSSc.

Objective: To determine the optimal treatment strategy in early dcSSc: the effect of HSCT as upfront therapy compared with that of immunosuppressive medication in early dcSSc, with respect to survival and prevention of major organ failure (referred to as 'event-free survival' which is considered as primary endpoint), safety and the impact on skin thickening, visceral involvement, functional status, and quality of life

Secondary goals are to evaluate (in both treatment arms) whether disease activity correlates with immunological parameters, including immunopathology of skin, immune reconstitution, and autoantibodies. We will also de-termine the cost-effectiveness of HSCT as first line treatment versus usual care and try to identify factors associated with response to treatment.

Study design: This investigation is an international multicentre, prospective, randomized, open label trial com-paring two treatment strategies used in regular care: upfront autologous HSCT versus immunosuppressive thera-py with i.v. CYC pulse therapy followed by MMF and HSCT as rescue option.

Study population: Patients aged between 18 - 65 years with an established diagnosis of dcSSc according to the ACR/EULAR criteria. Patients disease duration (non-Raynaud's symptoms) should be ≤ 3 years and mRSS ≥ 15 (diffuse skin pattern) and /or clinically significant organ involvement (heart and lung involvement).

Intervention: One group (A) receives upfront autologous HSCT and the other group (B) receives 12 monthly i.v. pulses CYC (750 mg/m2), followed by at least 12 months of oral MMF (max 3 grams daily) at one year after start of treatment. Rescue therapy may be considered in both arms in case of insufficient response or clinically relevant flare, but preferably not within the first 3 months after randomisation. For patients from Arm A methotrexate, mycophenolate mofetil or mycophenolic acid, or rituximab can be (re)instituted, according to local preference. Based on earlier studies, the clinical benefits of i.v. pulse cyclophosphamide may take between 6-12 months. Therefore it is recommended to then switch patients from arm B to HSCT only in case of rapidly progressive disease, which is arbitrarily defined as ≥30% increase in mRSS or ≥20% relative decline in FVC, TLC, or DLCO predicted.

Main study parameters/endpoints: Global Rank Composit score at 24 months follow-up.

Secondary efficacy endpoints: Event-free survival after randomisation/treatment, overall survival (OS), progression-free survival, number of participants that need rescue therapy (i.e. the alternative treatment) due to treatment failure. Treatment related mortality, treatment toxicity, and changes in mRSS, FVC, TLC and DLCO, nailfold microscopy, immunological markers in skin and blood, cardiac MR and 18FDG-PET. The CRISS at 12 months. Safety and tolerability outcomes according to CTC-criteria (CTCAE v5.0). Patient reported outcomes at 12 and 24 months include: Quality of life (EQ-5D), SHAQ, Gastrointestinal complaints (UCLA SCTC GIT 2.0), sexual functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years.
2. Fulfilling the 2013 ACR-EULAR classification criteria for SSc

   Either: 3.1 or 3.2 3.1. Disease duration ≤ 3 years (from onset of first non-Raynaud's symptoms) and diffuse cutaneous disease with

   - progressive skin involvement with a mRSS ≥ 15 (in a diffuse pattern: involvement of skin on the upper limbs, chest and/or abdomen)

   and/or

   - major organ involvement as defined by either:

   a. clinically significant respiratory involvement = i. DLCO and/or (F)VC ≤ 85% (of predicted) and evidence of interstitial lung disease on HR-CT scan with clinically relevant obstructive disease and emphysema excluded. ii. Patients with a DCLO and/or FVC > 85%, but with a progressive course of lung disease: defined as rela-tive decline of >10% in FVC predicted and/or TLC predicted, or >15% in DLCO predicted and evidence of interstitial lung disease on HR-CT scan with clinically relevant obstructive disease and emphysema ex-cluded, within 12 months. Intercurrent infections excluded.

   b. clinically significant renal involvement = i. new renal insufficiency (serum creatinine > upper limit of normal) AND
   1. persistent urinalysis abnormalities (proteinuria, haematuria, casts), AND/OR
   2. microangiopathic haemolytic anaemia AND/OR
   3. hypertension (two successive BP readings of either systolic ≥ 160 mm Hg or diastolic > 110 mm Hg, at least 12 hours apart), ; non-scleroderma related causes (e.g. medication, infection etc.) must be reasonably excluded.

   c. clinically significant cardiac involvement = any of the following criteria: i. reversible congestive heart failure, ii. atrial or ventricular rhythm disturbances such as atrial fibrillation or flutter, atrial paroxysmal tachycar-dia or ventricular tachycardia, 2nd or 3rd degree AV block, iii. pericardial effusion (not leading to hemodynamic problems), myocarditis; non-scleroderma related causes must have been reasonably excluded

   3.2. Disease duration ≤ 1 year (from onset of first non-Raynaud's symptoms) and diffuse cutaneous disease with mRSS ≥ 10 and
   1. High risk ANA for organ based disease: ATA or ARA positivity and/ or
   2. Acute phase response (ESR > 25 mm/h and/or CRP > 10.0 mg/L )

4. Written Informed consent

Exclusion Criteria:

1. Pregnancy or unwillingness to use adequate contraception during study
2. Concomitant severe disease =

   1. respiratory: resting mean pulmonary artery pressure (mPAP) > 25 mmHg (by right heart catheterisation), DLCO < 40% predicted, respiratory failure as defined by the primary endpoint
   2. renal: creatinine clearance < 40 ml/min (measured or estimated)
   3. cardiac: clinical evidence of refractory congestive heart failure; LVEF < 45% by cardiac echo or cardiac MR; chronic atrial fibrillation necessitating oral anticoagulation; uncontrolled ventricular arrhythmia; pericardial effusion with hemodynamic consequences
   4. liver failure as defined by a sustained 3-fold increase in serum transaminase or bilirubin, or a Child-Pugh score C
   5. psychiatric disorders including active drug or alcohol abuse
   6. concurrent neoplasms or myelodysplasia
   7. bone marrow insufficiency defined as leukocytopenia < 4.0 x 109/L, thrombocytopenia < 50x 10^9/L, anaemia < 8 gr/dL, CD4+ T lymphopenia < 200 x 106/L
   8. uncontrolled hypertension
   9. uncontrolled acute or chronic infection, including HIV, HTLV-1,2 positivity
   10. ZUBROD-ECOG-WHO Performance Status Scale > 2
3. Previous treatments with immunosuppressants > 12 months including MMF, methotrexate, azathioprine, rituximab, tocilizumab, glucocorticosteroids.
4. Previous treatments with TLI, TBI or alkylating agents including CYC.
5. Significant exposure to bleomycin, tainted rapeseed oil, vinyl chloride, trichlorethylene or silica;
6. eosinophilic myalgia syndrome; eosinophilic fasciitis.
7. Poor compliance of the patient as assessed by the referring physicians.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-17 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Global Rank Composite Score (GRCS) | 24 months
  The GRCS is an analytic tool that accounts for multiple disease manifestations simultaneously.
  For this endpoint, seveal endpoints will be used: death, event-free survival (EFS), forced vital capacity (FVC), Health Assessment Questionnaire - Disability Index (HAQ-DI), and Modified Rodnan Skin Score (mRSS).
  Participants alive ranked higher than those who died; those who survived event-free ranked higher than EFS failures. EFS failure included death, respiratory failure (decrease from baseline of >30% in DLCO % predicted or >20% in FVC % predicted ), renal failure (chronic dialysis > 6 month or renal transplant), or cardiac failure (clinical congestive heart failure or left ventricular ejection fraction <30%). The lowest 3 GRCS components are ordinal; improvement, stability, or worsening from baseline (±10% change in FVC % predicted, ±0.4 change in HAQ-DI, ±25% change in mRSS).

SECONDARY OUTCOMES:
Number of patients who survive without disease progression (Progression-free survival) | 24 months
  Defined as the time in days since the day of randomisation until any of the following relative changes from base-line has been documented:
  * death,
  * ≥ 10% drop in (F)VC predicted and/or ≥ 15% drop in DLCO predicted,
  * ≥ 15% drop in LVEF by echo or cardiac MR,
  * ≥ 15% drop in body weight,
  * ≥ 30% drop in creatinine clearance,
  * ≥ 30% increase in skin score,
  * ≥ 0.5 increase in SHAQ.
Number of patients who die due to complications related to the treatment (Treatment related mortality) | 24 months
  Defined as any death during the study period following randomisation that cannot be attributed to progression of the disease according to the consensus opinion of the DSMB.
Number of patient alive after 24 months (Overall mortality) | 24 months
  Any death, regardless of relationship to treatment, between randomization and 24 months post-randomization
Number of CTCAE toxicity advserse events | 24 months
  Number of CTCAE v5.0 toxicity advserse events =/> grade 3 that occur in consecutive 3-month periods following randomisation until 24 months follow-up.
The area under the curve (AUC) of the CRISS over time | 24 months
  The American College of Rheumatology Composite Response Index in Diffuse Cutaneous Systemic Sclerosis (ACR CRISS) was developed using expert consensus and data driven approaches for use in clinical trials (Khanna et al, 2016).
  The exponential algorithm determines the predicted probability of improvement from baseline, incorporating change in the mRSS, FVC percent predicted, physician and patient global assessments, and HAQ-DI. The outcome is a continuous variable between 0.0 and 1.0 (0 - 100%). A higher score indicates greater improvement. Subjects are not considered improved (ACR CRISS score = 0) if they develop new: 1) renal crisis; 2) decline in FVC% predicted by 15% (relative) from baseline and confirmed after 1 month; or 3) left ventricular failure (systolic ejection fraction < 45%); or 4) new pulmonary artery hypertension on right heart catheterization requiring treatment.
Changes in skin involvement (modified Rodnan Skin Score) | 24 months
  Modified Rodnan Skin Score (mRSS) The MRSS is a validated physical examination method for estimating skin induration. It is correlated with biopsy measures of skin thickness and reflects prognosis and visceral involvement, especially in early disease2, 4. It is scored on a 0 (normal) to 3+ (severe induration) ordinal scales over 17 body areas, with a maximum score of 51 and is used to categorize severity of SSc. Minimally clinically significant difference in MRSS is 3-5 points (Amjadi et al., American College of Rheumatology; Aug 2009; 2493-2494) It has been extensively used as primary/ secondary outcome in RCT with Scleroderma. This will be collected at every study visit.
Changes in cardiac function(Left Ventricular Ejection Fraction) | 12 and 24 months
  LVEF is measured by cardiac echo and at baseline and 12 months with cardiac MRI.
Changes in pulmonary function | 12 and 24 months
  Diffusion in liters of carbon monoxide (DLCO) is a measure of lung function. Predicted values for DLCO were computed using the Crapo Morris equations and adjusted per the Cotes formula for anemia, if a participant's hemoglobin was <13 or >17 gm/dL, and altitude (Calgary site only). Forced Vital Capacity (FVC) is the amount of air that can be forcibly exhaled after a full breath and is a measure of lung function. Predicted FVC was based on institutional standards.
Changes in health related quality of life EQ-5D-5L index | 24 months
  HR-QoL will be assessed using the validated EuroQol (EQ-5D-5L), the calculated index ranges from 0 (worse HR-QoL) to 1 (best HR-QoL).
Changes in nailfold capillaroscopy | 12 and 24 months
  Nailfold capillaroscopy (NFS) will be obtained by the local capillaroscopist pre- and post-ASCT (at baseline, at 6, 12 24 months and yearly after). The evaluation of the images will be done centrally. The NFS-findings will be described standardly according to the consensus of the EULAR study group on microcirculation in rheumatic diseases. As such, the images will be evaluated in a quantitative (density, di-mension, morphology and presence of haemorrhages) and a qualitative way (normal, aspecific abnormalities, early/active/late scleroderma pattern). As we will analyse 16 NFS-images per subject, an overall qualitative as-sessment per subject will be assigned, based on the most prevalent pattern per subject.
Changes in 18F FDG-PET scan from the thorax | 12 months
  Validation of semi-quantitative analysis method with respiratory gated and non-gated 18F FDG-PET prospec-tively and comparison of 18F FDG-PET with routine HR-CT thorax, pulmonary lung function and clinical symptoms, will be done at baseline and at 12 months follow-up.
Changes in gastrointestinal complaints (UCLA SCTC GIT 2.0) | 12 and 24 months
  The UCLA SCTC GIT 2.0 is a standardized set of outcome measures developed through literature review, patient focus groups and cognitive debriefing among patients with a variety of gastrointestinal disorders including irritable bowel syndrome, inflammatory bowel disease, other common gastrointestinal disorders, SSc, and a census-based US general population control sample (Khanna et al, 2009). The scale consists of eight domains relating to gastroesophageal reflux (13 items), disrupted swallowing (7 items), diarrhea (5 items), bowel incontinence/soilage (4 items), nausea and vomiting (4 items), constipation (9 items), belly pain (6 items), and gas/bloat/flatulence (12 items). The scales correlated significantly with both generic and disease-targeted legacy instruments, and demonstrate evidence of reliability.
Changes in several subsets of the immune system | 12 months
  We will evaluate antibody repertoire pre- and post-treatment at dedicated timepoints and assess correlations to clinical disease course characteristics. Also, B cells will be characterized in terms of frequency, phenotype and functional capacities before and after treatment. Additionally, transcriptomics analysis on the immune cell (sub-)populations isolated will be done.
Changes in self-assessed skin thickness (PASTUL_) | 60 months
  Patients will assess their skin thickness using the validate PASTUL questionnaire every 3 months.
Inflammatory and fibrotic characteristics and changes of the skin and composition of the microbiome of the skin | 12 months
  Skin biopsies from affected skin will be used to investigate the inflammatory and fibrotic changes and the skin microbiome. Before taking the skin biopsies the skin will be anesthetized with lidocaine 1%. The biopsy used for analysis of the inflammatory and fibrotic characteristics, using immunohistochemistry, will be frozen in liquid nitrogen. 6S rRNA gene sequencing will be done to obtain the microbial profiles of the skin biopsies.
Changes in sexual functioning | 12 and 24 months
  We will use the validated IIEF-5 and SFQ-28
Changes in daily functioning | 12 and 24 months
  SHAQ-DI The SHAQ-DI is a disease-targeted, musculoskeletal-targeted measure intended for assessing functional ability in scleroderma. It is a self-administered 20-question instrument that assesses a patient's level of functional ability and includes questions that involve both upper and lower extremities. The SHAQ-DI score ranges from 0 (no disability) to 3 (severe disability). It has a 7 day recall period and has been extensively used in SSc. Five visual analog scales are included in the scleroderma-HAQ assessing burden of digital ulcers, Raynaud's, gastrointestinal involvement, breathing, and overall disease.
Changes in ability to work, measured by the customized Productivity Cost Questionnaire (iPCQ) | 12 and 24 months
  The customized iPCQ is a selection of 5 questions derived from the full iPCQ
Changes in fatigue measured with the FACIT questionnaire | 12 and 24 months
  The FACIT questionnaire is a validated questionnaire for evaluating fatigue
Changes in handmobility | 24 months
  assessment done using the mHAMIS
Number of patients who survive without major events (event free survival) | 24 months
  Event-free survival is defined as the time in days from the day of randomisation until the occurrence of death due to any cause or the development of persistent major organ failure (heart, lung, kidney) defined as follows:
  * Heart: left ventricular ejection fraction < 30% by cardiac MR (or cardiac echo)
  * Lungs: respiratory failure = resting arterial oxygen tension (PaO2) < 8 kPa (< 60 mmHg) and/or resting arterial carbon dioxide tension (PaCO2) > 6.7 kPa (> 50 mmHg) without oxygen supply
  * Kidney: need for renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jacob M van Laar, MD PhD, Principal Investigator — UMC Utrecht; Julia Spierings, Study Director — UMC Utrecht
Locations (12):
- Italy (3):
  - Gaetano Pini-CTO, Milan
  - Ospedale San Raffaele, Milan
  - University Hospital Rome, Roma
- Netherlands (4):
  - Amsterdam Rheumatology Centre, Amsterdam
  - University Medical Centre Leiden, Leiden
  - Radboudumc Nijmegen, Nijmegen
  - University Medical Centre Utrecht, Utrecht
- Sweden (2):
  - Skåne University Hospital Lund, Lund
  - Karolinska Institute/Karolinska University Hospital Solna, Stockholm
- Switzerland (2):
  - University Hospital Basel, Basel
  - Inselspital, Universitätsspital Bern, Bern
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Burt RK, Shah SJ, Dill K, Grant T, Gheorghiade M, Schroeder J, Craig R, Hirano I, Marshall K, Ruderman E, Jovanovic B, Milanetti F, Jain S, Boyce K, Morgan A, Carr J, Barr W. Autologous non-myeloablative haemopoietic stem-cell transplantation compared with pulse cyclophosphamide once per month for systemic sclerosis (ASSIST): an open-label, randomised phase 2 trial. Lancet. 2011 Aug 6;378(9790):498-506. doi: 10.1016/S0140-6736(11)60982-3. Epub 2011 Jul 21. PMID 21777972
- [Background] Sullivan KM, Goldmuntz EA, Keyes-Elstein L, McSweeney PA, Pinckney A, Welch B, Mayes MD, Nash RA, Crofford LJ, Eggleston B, Castina S, Griffith LM, Goldstein JS, Wallace D, Craciunescu O, Khanna D, Folz RJ, Goldin J, St Clair EW, Seibold JR, Phillips K, Mineishi S, Simms RW, Ballen K, Wener MH, Georges GE, Heimfeld S, Hosing C, Forman S, Kafaja S, Silver RM, Griffing L, Storek J, LeClercq S, Brasington R, Csuka ME, Bredeson C, Keever-Taylor C, Domsic RT, Kahaleh MB, Medsger T, Furst DE; SCOT Study Investigators. Myeloablative Autologous Stem-Cell Transplantation for Severe Scleroderma. N Engl J Med. 2018 Jan 4;378(1):35-47. doi: 10.1056/nejmoa1703327. PMID 29298160
- [Background] van Laar JM, Farge D, Sont JK, Naraghi K, Marjanovic Z, Larghero J, Schuerwegh AJ, Marijt EW, Vonk MC, Schattenberg AV, Matucci-Cerinic M, Voskuyl AE, van de Loosdrecht AA, Daikeler T, Kotter I, Schmalzing M, Martin T, Lioure B, Weiner SM, Kreuter A, Deligny C, Durand JM, Emery P, Machold KP, Sarrot-Reynauld F, Warnatz K, Adoue DF, Constans J, Tony HP, Del Papa N, Fassas A, Himsel A, Launay D, Lo Monaco A, Philippe P, Quere I, Rich E, Westhovens R, Griffiths B, Saccardi R, van den Hoogen FH, Fibbe WE, Socie G, Gratwohl A, Tyndall A; EBMT/EULAR Scleroderma Study Group. Autologous hematopoietic stem cell transplantation vs intravenous pulse cyclophosphamide in diffuse cutaneous systemic sclerosis: a randomized clinical trial. JAMA. 2014 Jun 25;311(24):2490-8. doi: 10.1001/jama.2014.6368. PMID 25058083
- [Background] van Bijnen S, de Vries-Bouwstra J, van den Ende CH, Boonstra M, Kroft L, Geurts B, Snoeren M, Schouffoer A, Spierings J, van Laar JM, Huizinga TW, Voskuyl A, Marijt E, van der Velden W, van den Hoogen FH, Vonk MC. Predictive factors for treatment-related mortality and major adverse events after autologous haematopoietic stem cell transplantation for systemic sclerosis: results of a long-term follow-up multicentre study. Ann Rheum Dis. 2020 Aug;79(8):1084-1089. doi: 10.1136/annrheumdis-2020-217058. Epub 2020 May 14. PMID 32409324
- [Derived] Spierings J, van Rhenen A, Welsing PM, Marijnissen AC, De Langhe E, Del Papa N, Dierickx D, Gheorghe KR, Henes J, Hesselstrand R, Kerre T, Ljungman P, van de Loosdrecht AA, Marijt EW, Mayer M, Schmalzing M, Schroers R, Smith V, Voll RE, Vonk MC, Voskuyl AE, de Vries-Bouwstra JK, Walker UA, Wuttge DM, van Laar JM. A randomised, open-label trial to assess the optimal treatment strategy in early diffuse cutaneous systemic sclerosis: the UPSIDE study protocol. BMJ Open. 2021 Mar 18;11(3):e044483. doi: 10.1136/bmjopen-2020-044483. PMID 33737437
- See also: official trial website — http://upsidetrial.com/